CLINICAL TRIAL: NCT06582316
Title: Digital Solution for Salutogenic Brain Health (DiSaB): A Pilot Sequential Multiple Assignment Randomised Trial (SMART) Protocol for Clinical Implementation
Brief Title: Digital Solution for Salutogenic Brain Health (DiSaB): A Pilot Protocol for Clinical Implementation
Acronym: DiSaB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Catherine Yanhong Dong, PhD, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023/00620
Record Dates: First submitted 2024-08-16; First posted 2024-09-03 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-08

CONDITIONS: Chronic Condition
Keywords: Cognition; Implementation Science; Digital Intervention; Hypertension; Hyperlipidaemia; Type-2 Diabetes
MeSH Terms: conditions — Chronic Disease; Hypertension; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Participants will undergo 8 sessions of digital "Train Your Brain" programme lead by a trained clinical neuropsychologist over 2 months.
  Interventions: Other: Brain Health Training Programme
- Control Arm (No Intervention): Participants will not undergo any sessions of digital "Train Your Brain" programme for 2 months when intervention arm's brain health training programme is ongoing.

INTERVENTIONS:
Other: Brain Health Training Programme — "Train Your Brain (TYB)" - group-based cognitive intervention programme for mild cognitive impairments. This programme equips participants with knowledge on cognition and brain health, provide cognitive coping strategies and boost their confidence and maintain independence in daily activities.
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to develop and learn if a digitally delivered brain health intervention (DiSaB) can help improve cognitive, physical and psychosocial health in middle-aged adults with chronic conditions at-risk for cognitive decline. The clinical trial also aims to find out the push and pull factors of implementing the intervention in primary care settings. The main questions it aims to answer are:

1. Does the DiSaB intervention improve participants' cognitive functions, health measures, and psychosocial health?
2. Is an individualised or group-based health education session better at improving cognitive, physical and psychosocial health in participants who did not respond to the DiSaB intervention?
3. How useful and practical is the DiSaB intervention, according to

   1. participants and
   2. nurses carrying out the intervention?

The investigators will compare a DiSaB intervention to a control condition (where participants do not undergo any intervention) to see if the DiSaB intervention works in improving participants' health.

The investigators will also compare individualised versus group health education sessions to see which session is better at improving the health of participants who did not respond to the DiSaB intervention.

Participants will

1. Complete cognitive assessments, questionnaires, and health tests before intervention, immediately after the intervention, and 6 months after the intervention
2. Either undergo no intervention, or undergo the DiSaB intervention over 2 months
3. Be randomly selected to attend focus group interviews

Local champions will complete questionnaires and attend focus group interviews after administering and/or co-facilitating the intervention.

DETAILED DESCRIPTION:
The effectiveness of the DiSaB intervention implementation at primary care setting amongst participants with long term conditions will be evaluated using the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) model.

Secondly, the barriers and facilitators to DiSaB implementation amongst local champions [e.g., advanced practice nurses (APNs)] will be determined. Specifically, using the Capability, Opportunity, Motivation and Behavior (COM-B) model, the investigators will evaluate the barriers and facilitators towards DiSaB intervention implementation among healthcare professionals.

Third, sequential multiple assignment randomised trial (SMART) study design will also be employed in this study for the development of dynamic treatment regimens (DTRs) tailored for individual needs. The investigators first aim to evaluate the feasibility and compare the efficacy of additional individual intervention (i.e. a health education individual feedback session within 1 - 2 months) vs a smaller group intervention (i.e. health education group sessions over 3 months, once per month) post-standard TYB intervention amongst non-responders, in improving cognitive functions and management of their long-term conditions. Finally, the investigators will compare two embedded DTRs in the SMART, namely, (1) standard TYB followed by individualised health education session for non-responders and usual care for responders, and (2) standard TYB followed by group health education session for non-responders and usual care for responders.

Lastly, an economic evaluation will be carried out to evaluate cost-effectiveness and further impacts of the DiSaB implementation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 - 55 years old
* Have hypertension, hyperlipidaemia and/or type-2 diabetes
* Ability to provide written informed consent
* Posses sufficient English language skills in reading, writing and speaking
* Multimorbidity conditions are also acceptable with the exception of life-threatening co-morbidities with life expectancy of less than one year
* Total Risk Score (TRS) for cognitive impairment of at least 3

Exclusion Criteria:

* Physical, visual and/or hearing impairment
* Language impairment (i.e. severe dysarthria or aphasia)
* Not within age range listed
* Major or active psychiatric conditions
* Diagnosis of dementia
* Do not own a mobile device capable of downloading applications (i.e. Zoom), and/or do not have access to internet connection

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate | Baseline (all participants; month 0), first follow up (all participants; month 3), second follow up (only for control group; at month 6), and final follow up (all participants; months 9/12)
  Heart rate will be measured on-site
Change in lipid levels | Baseline (all participants; month 0), first follow up (all participants; month 3), second follow up (only for control group; at month 6), and final follow up (all participants; months 9/12)
  Information will be obtained from patients; HealthHub/Health Buddy/OneNUHS or other health apps
Change in HbA1c levels | Baseline (all participants; month 0), first follow up (all participants; month 3), second follow up (only for control group; at month 6), and final follow up (all participants; month 9/12)
  Information will be obtained from patients; HealthHub/Health Buddy/OneNUHS or other health apps
Change in blood pressure | Baseline (all participants; month 0), first follow up (all participants; month 3), second follow up (only for control group; at month 6), and final follow up (all participants; month 9/12)
  Blood pressure will be measured on-site
Change in SDMT scores | Baseline (all participants; month 0), first follow up (all participants; month 3), second follow up (only for control group; at month 6), and final follow up (all participants; month 9/12)
  Symbol Digit Modality Test (SDMT). Total maximum score is 110. Higher scores indicate better cognitive performance.
Change in psychosocial health measured by DaSS-21 | Baseline (all participants; month 0), first follow up (all participants; month 3), second follow up (only for control group; at month 6), and final follow up (all participants; month 9/12)
  Depression, Anxiety and Stress Scale -21 item (DASS-21) Physical or online. There are 21 questions that are scored from 0 to 3, and the highest possible score is 63. Higher scores indicate poorer psychological health.
Change in MoCA scores | Baseline (all participants; month 0), first follow up (all participants; month 3), second follow up (only for control group; at month 6), and final follow up (all participants; month 9/12)
  Montreal Cognitive Assessment (MoCA). Total possible score is 30 (scoring is on the MoCA form itself), and a score of at least 26 indicates normal cognition. Higher scores indicate better cognition.
Change in quality of life measured by EQ-5D-5L | Baseline (all participants; month 0), first follow up (all participants; month 3), second follow up (only for control group; at month 6), and final follow up (all participants; month 9/12)
  EuroQol 5 Dimension 5 Level (EQ-5D-5L) Physical or online. Each question is scored from 1 to 5, with 1 indicating no problems in that dimension and 5 indicating total inability to perform in that dimension.
Change in psychosocial health measured by AD8 | Baseline (all participants; month 0), first follow up (all participants; month 3), second follow up (only for control group; at month 6), and final follow up (all participants; month 9/12)
  Alzheimer's Disease-8 Component (AD8) Physical or online. There are a total of 8 questions asking about thinking ability, and each answer is coded 1 (yes, change present) or 0 (no change). 0 or 1 indicates normal cognition, and a score of at least 2 suggests that cognition issues might be present.
Change in psychosocial health measured by Self-care of chronic illness inventory | Baseline (all participants; month 0), first follow up (all participants; month 3), second follow up (only for control group; at month 6), and final follow up (all participants; month 9/12)
  Physical or online. 29 questions in total, answers are scored from 1 to 5. Higher scores indicate better self-care. When referencing standard scores, a standard score of 70 is the cut-off point for self-care adequacy.
Patient satisfaction feedback questionnaire (patients) | Weekly (right after each TYB intervention) for 2 months. Also after health education sessions: either once [individual session] OR monthly for 3 months [group session]; during months 4-6) - intervention arm non-responders only
  Completed online
Feedback from patients using focus group interview | Final follow up (month 9/12)
  Questions are developed from RE-AIM model. Participants will be randomly chosen (n=30) to take part in the focus group interview.
Effectiveness of TYB intervention questionnaire (nurses) | Weekly for 2 months (after each TYB intervention - months 1-3 for intervention arm and months 4-6 for control arm), final follow up (month 12)
  Using RE-AIM model; completed online. Questionnaire will be given at multiple time points throughout the study, as listed below.
Effectiveness of DiSaB intervention questionnaire (patients) | Once at the end of TYB intervention (month 3 for intervention arm, month 6 for control arm), once during final follow-up (month 9/12 for all participants)
  Using RE-AIM model; completed online. Questionnaire is given at multiple points throughout the study, as listed below.
Feedback from nurses using focus group interview | Month 6 (immediately after completion of 2-month-long TYB intervention control arm)
  Questions are developed from RE-AIM model

SECONDARY OUTCOMES:
Economic evaluation on the feasibility of DiSaB implementation using cost-effectiveness questionnaire | Baseline (all participants; month 0), first follow up (all participants; month 3), second follow up (only for control group; at month 6), and final follow up (all participants; months 9/12)
  For evaluation of economics and further impact

CONTACTS AND LOCATIONS:
Locations (1):
- National University Polyclinics, Singapore, Singapore

REFERENCES:
- [Derived] Chang CSY, Phua V, Tham XC, Jia Y, Chen NYC, Zhou W, Liau WF, Xu J, Chakraborty B, Graves N, Sevdalis N, Dong Y. Digital solution for salutogenic brain health: a pilot sequential multiple assignment randomised trial (SMART) protocol for clinical implementation. BMJ Open. 2025 Mar 25;15(3):e096568. doi: 10.1136/bmjopen-2024-096568. PMID 40132849